CLINICAL TRIAL: NCT03254017
Title: Remotely Programmed Deep Brain Stimulation of the Bilateral Habenula for Treatment- Resistant Major Depression: An Open Label Pilot Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: logistics reasons
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Bomin Sun, Director of the Department of Functional Neurosurgery, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Habenula DBS
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Treatment Resistant Major Depressive Disorder
Keywords: Bilateral Habeluna; Remote Deep Brain Stimulation; Treatment Resistant Major Depressive Disorder

STUDY DESIGN:
Intervention Model Description: all subjects will receive bilateral surgical implantation of DBS system.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Deep Brain Stimulation (Experimental): Device：Suzhou Sceneray® DBS system
  Interventions: Procedure: Bilateral surgical implantation of DBS system to Habeluna; Other: Follow-up Period

INTERVENTIONS:
Procedure: Bilateral surgical implantation of DBS system to Habeluna — The SceneRay DBS device utilized in the present study is a double-channel device designed and manufactured by Suzhou Scene-Ray Medical Co., Ltd. The DBS system includes a dual-channel neurostimulator kit, lead kit, extension kit, clinician-operated wireless programmer, test stimulator, and patient controller. The lead (diameter =1.27 mm) contains four stimulating contacts made of platinumiridium alloy. The length of each contact is 1.5 mm, and interval spaces are 0.5 mm. This device shares the same basic principles utilized by Medtronic products, with unique wireless programming and electrode fixing designs. The amplitude (0-10 V), pulse width (60-960 ms), and frequency (1-1,600 Hz) can be programmed, and different frequencies may be utilized in the left and right hemispheres using this type of dual-channel IPG.
Other: Follow-up Period — The researchers will remotely program the DBS biweekly after opening the stimulator and face to face test the patients' cognitive function every half year. Montgomery-Asberg Depression Rating Scale will be tested biweekly until the Programmed parameter has stable therapeutic efficacy and then tested after 3 months, 6 months, 9 months and 12 months.The other neuropsychological scales will be test on 3 months, 6 months, 9 months and 12 months.

SUMMARY:
The habenula(Hb) is an epithalamic structure located at the center of the dorsal diencephalic conduction system, a pathway involved in linking forebrain to midbrain regions. An increasing number of studies indicates that that overactivity in the lateral habeluna(LHb) is present during depressed states, where it could drive the changes in midbrain activity linked to depression. Deep brain stimulation(DBS) of the major afferent bundle (i.e., stria medullaris thalami) of the LHb can treat treatment-resistant major depression(TRD). There is no clinical case of directly stimulating habeluna for treatment TRD. This research will investigate effectiveness bilateral DBS to habenula for patients with TRD.

Programming is a crucial aspect of DBS which directly influences its therapeutic efficacy. Researchers need to ascertain optimum stimulation parameters to help patients achieve optimal control of clinical symptoms. Remote programming of DBS can markedly improve patient convenience, minimize risk of infection and total treatment time and lead to an overall benefit for doctors and patients alike. This research will also investigate safety and benefit of remote programming of DBS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old
* Proficiency in Mandarin language;
* DSM-IV diagnosis of Majior depression disorder;
* Current episode duration ≥ 2 years;
* Failure to respond to a minimum of four different antidepressant treatments;
* Failure or intolerance of an adequate course of electroconvulsive therapy (ECT) during any episode;
* Capacity to provide informed consent (understanding of the study purpose and methods);

Exclusion Criteria:

* Schizophrenia or history of psychosis unrelated to MDD;
* Antisocial personality disorder, dementia, current tic disorder;
* Past stereotactic neurosurgical intervention;
* Alcohol or substance abuse/dependence within 6 months;
* Neurological disease (Abnormal PET-CT, MRI, EEG);
* Contraindications of MRI-examination, e.g. implanted cardiac pacemaker/ heart defibrillator;
* Contraindications of stereotactic intervention, e.g. increased bleeding disposition, cerebrovascular diseases;
* Serious and unstable organic diseases (e.g. unstable coronal heart disease);
* HIV positive;
* Pregnancy and/or lactation;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Change in the Montgomery-Asberg Depression Rating Scale | Baseline (preoperative),Biweekly after onset of the DBS system,3 months,6 months, 9 months, 12 months
Change in the Hamilton Depression Scale | Baseline（preoperative）,3 months, 6 months,9 months, 12months

SECONDARY OUTCOMES:
Change in the Hamilton Anxiety Scale | Baseline（preoperative）,3 months, 6 months,9 months, 12months
Change in the Quality of Life Assessment (SF-36) | Baseline（preoperative）,3 months, 6 months,9 months, 12 months
Neuropsychological measures(Scores of cogstate battery) | Baseline（preoperative）,6 months,12 months
Change in the Hamilton Anxiety Scale | Baseline（preoperative）,3 months, 6 months,9 months, 12 months
Change in the WHO-BREF | Baseline（preoperative）,3 months,6 months,9 months, 12 months
Change in Young Manic Rating Scale | Baseline (preoperative),Biweekly after onset of the DBS system,3 months,6 months, 9 months, 12 months
Chang in Pittsburgh Sleep Quality Index | Baseline（preoperative）,3 months,6 months,9 months, 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ruijin Hospital Functional Neurosurgery, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Sartorius A, Kiening KL, Kirsch P, von Gall CC, Haberkorn U, Unterberg AW, Henn FA, Meyer-Lindenberg A. Remission of major depression under deep brain stimulation of the lateral habenula in a therapy-refractory patient. Biol Psychiatry. 2010 Jan 15;67(2):e9-e11. doi: 10.1016/j.biopsych.2009.08.027. No abstract available. PMID 19846068
- [Background] Kiening K, Sartorius A. A new translational target for deep brain stimulation to treat depression. EMBO Mol Med. 2013 Aug;5(8):1151-3. doi: 10.1002/emmm.201302947. Epub 2013 Jul 4. No abstract available. PMID 23828711
- [Background] Fakhoury M. The habenula in psychiatric disorders: More than three decades of translational investigation. Neurosci Biobehav Rev. 2017 Dec;83:721-735. doi: 10.1016/j.neubiorev.2017.02.010. Epub 2017 Feb 13. PMID 28223096
- [Background] Proulx CD, Hikosaka O, Malinow R. Reward processing by the lateral habenula in normal and depressive behaviors. Nat Neurosci. 2014 Sep;17(9):1146-52. doi: 10.1038/nn.3779. PMID 25157511
- [Background] Bergfeld IO, Mantione M, Hoogendoorn ML, Ruhe HG, Notten P, van Laarhoven J, Visser I, Figee M, de Kwaasteniet BP, Horst F, Schene AH, van den Munckhof P, Beute G, Schuurman R, Denys D. Deep Brain Stimulation of the Ventral Anterior Limb of the Internal Capsule for Treatment-Resistant Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2016 May 1;73(5):456-64. doi: 10.1001/jamapsychiatry.2016.0152. PMID 27049915
- [Background] Li D, Zhang C, Gault J, Wang W, Liu J, Shao M, Zhao Y, Zeljic K, Gao G, Sun B. Remotely Programmed Deep Brain Stimulation of the Bilateral Subthalamic Nucleus for the Treatment of Primary Parkinson Disease: A Randomized Controlled Trial Investigating the Safety and Efficacy of a Novel Deep Brain Stimulation System. Stereotact Funct Neurosurg. 2017;95(3):174-182. doi: 10.1159/000475765. Epub 2017 Jun 2. PMID 28571034
- [Background] Zhang C, Li D, Zeljic K, Tan H, Ning Y, Sun B. A Remote and Wireless Deep Brain Stimulation Programming System. Neuromodulation. 2016 Jun;19(4):437-9. doi: 10.1111/ner.12448. No abstract available. PMID 27321195